CLINICAL TRIAL: NCT00715975
Title: Clinical Trial of Effectiveness and Safety of Topical Halobetasol Propionate in the Treatment of Patients With Psoriasis Plate, and as Comparator the Product Psorex (Clobetasol Propionate).
Brief Title: Effectiveness and Safety of Topical Halobetasol Propionate in the Treatment of Patients With Psoriasis
Acronym: halobetasol
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HALGLE0508
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-08

CONDITIONS: Psoriasis
Keywords: clobetasol; halobetasol; psoriasis; evaluating the efficacy and tolerability of the drug Halobetasol propionate
MeSH Terms: conditions — Psoriasis | interventions — halobetasol; Clobetasol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The patients will be treated with halobetasol once a day for 15 days.
  Interventions: Drug: halobetasol
- 2 (Experimental): The patients will be treated with clobetasol once a day for 15 days.
  Interventions: Drug: clobetasol

INTERVENTIONS:
Drug: halobetasol — The patients will be treated with halobetasol once a day for 15 days.
  Arms: 1
Drug: clobetasol — The patients will be treated with clobetasol once a day for 15 days.
  Arms: 2

SUMMARY:
The Psoriasis and a chronic dermatosis characterized by abnormal proliferation of cells epithelial, vessel dilation and inflammation locally, which presents erythematous-scaly lesions in various areas of the body, preferably in the scalp, region and religious joints as elbows and knees. It occurs equally in both sexes and can appear at any age, and the mean age for the onset of the disease and around 27.3 years.

The halobetasol propionate and an ultra-potent corticoid. Its chemical structure and similar to the Clobetasol corticoid this, until then classified as the most potent corticoid used worldwide in clinical practice. However, the molecular structure of Halobetasol gives it increased its activity antiinflammatory and anti-proliferative.

The objective of this study is evaluating the efficacy and tolerability of the drug Halobetasol propionate cream formulation as a treatment in patients with plaque psoriasis mild to moderate, compared to the substance of similar power, Clobetasol propionate - Psorex - Cream.

DETAILED DESCRIPTION:
The patients eligible will be informed about the procedures of the study and that agree to participate and sign the TCLE will be initially evaluated clinically for the clinical diagnosis of psoriasis plate with mild and moderate involvement of up to 20% of body surface. After the procedures for selection (initial clinical evaluation and verification of the criteria for inclusion and exclusion) the patients will be photographed, receive treatment and will be targeted and to manage it in proper way and standardized, when they do so at home. In each return (after 7, 14 days) will be held photographs of injuries, clinical examination, evaluation of adverse events and dispensing of medicine to patients.

The drugs dispensed will be sufficient for daily use until the next return. The product will be applied once a day, during night, preferably after the bath. The follow-up visits will occur in times of 07 and 14 days after the start of treatment. If there is complete improves the disease, treatment is interrupted before this date. On each visit will be examined by clinical parameters validated scales of assessment internationally (PASI), which provide the exact data of changes in the framework of each patient in each parameter measured. As parameters of the tolerability will be evaluated frequency and intensity of adverse events and the potential of irritative formulations, will be held photo of patients and questionnaires of cosmeticidade the formulation. Patients will be geared not to expose to the sun during the treatment period. At the end of the study, patients who present evolution will be full of injuries released the study and those who are still with obvious symptoms have treatment interrupted because of the risk of prolonged use of the drug under study. These patients will be referred to the Health Service for maintenance treatment with a new therapy. The patients who are released and make recurrence of the disease due to the rebound effect will be

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, adults over 18 years, holders of psoriasis plating of mild to moderate,
* Patients with area of involvement of up to 20% of body surface,
* Patients with good physical and mental health
* Patients who agree with the purposes of the study and sign the Informed Consent

Exclusion Criteria:

* Patients with skin diseases other than psoriasis or which alter the clinical evaluation and development of disease,
* Patients with psoriasis in more than 20% of the body,
* Patients with other types of psoriasis that are not "plating",
* patient with a scalp psoriasis who have difficulty in application of the product,
* Patients who have made topical treatment for psoriasis in the 2 months preceding the study,
* Patients who have made systemic treatment for psoriasis in the 4 months preceding the study,
* Patients who do not agree with the conditions described in the Statement of Informed Consent
* Patients who are pregnant and breastfeeding,
* Patients in use of oral anticoagulants,
* Patients who have psoriatics addition to plaques of skin disorders caused by fungi or bacteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
assess the improvement of symptoms of psoriasis | complete improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica, Valinhos, São Paulo, Brazil